CLINICAL TRIAL: NCT03285633
Title: Telephone-Based Mindfulness CBT for Patients in Community Settings With Advanced Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Palliative Care Research Cooperative Group (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00080262
Record Dates: First submitted 2017-09-14; First posted 2017-09-18 (Actual); Last update posted 2019-08-19 (Actual); Status verified 2019-08

CONDITIONS: Advanced Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cognitive Behavioral Mutli-Symptom management(CBT) (Other): Learn to manage distress, fatigue, and/or pain via Cognitive Behavioral Multi-Symptom Management(CBT). Four sessions will be conducted each session is approximately one hour.
  Interventions: Behavioral: Cognitive Behavioral Mutli-Symptom management(CBT)

INTERVENTIONS:
Behavioral: Cognitive Behavioral Mutli-Symptom management(CBT) — Learn to manage distress, fatigue, and/or pain via (Cognitive Behavioral Multi-Symptom management (CBT) four one hour sessions.

SUMMARY:
This study examines the feasibility and acceptability of an open trial of mindfulness-based Cognitive Behavioral Therapy intervention delivered via telephone to men and women age 21 and older with a diagnosis of advanced cancer. Potential participants (N=35) will be recruited via letter from their oncologist at community-based clinics (N=18) and those served at the Duke Cancer Institute in Durham who live more than 60 miles away (N=17). Following informed consent, participants will be asked to complete assessments (e..g., examining their pain, anxiety, depression, fatigue, and engagement in valued activity). They will then receive 4 weekly 50-minute telephone sessions with a study therapist and practice skills learned in session at home. After completing the 4 sessions, they will complete a post-treatment assessment. Data analyses will examine the feasibility and acceptability of the study by assessing participant engagement, and will examine changes in key psychological variables (e.g., pain, anxiety, depression, fatigue, and valued activity) from baseline to post-treatment.

DETAILED DESCRIPTION:
Individuals with advanced cancers often experience significant symptom burden including pain, fatigue, and psychological distress, all while facing acceptance of the meaning of their advanced disease. Evidence-based behavioral interventions have been developed to alleviate this multiple symptom burden but are understudied and the treatments that are available are often not easily accessed by patients most in need in community-based settings. The current study examines the feasibility and acceptability of an open trial of mindfulness-based Cognitive Behavioral Therapy intervention delivered via telephone to men and women age 21 and older with a diagnosis of advanced cancer. Potential participants (N=35) will be recruited via letter from their oncologist at community-based clinics (N=18) and those served at the Duke Cancer Institute in Durham who live more than 60 miles away (N=17). Following informed consent, participants will be asked to complete assessments (e..g., examining their pain, anxiety, depression, fatigue, and engagement in valued activity). They will then receive 4 weekly 50-minute telephone sessions with a study therapist and practice skills learned in session at home. After completing the 4 sessions, they will complete a post-treatment assessment. Data analyses will examine the feasibility and acceptability of the study by assessing participant engagement, and will examine changes in key psychological variables (e.g., pain, anxiety, depression, fatigue, and valued activity) from baseline to post-treatment. There is minimal risk related to confidentiality of data and the possibility of feeling uncomfortable in the study. All study contacts will be conducted by trained study staff and supervised by the PI; a licensed clinical psychologist. Participant tracking data will be stored online via REDCAP and accessed only by study staff, participant assessment data will be collected and stored online via REDCap, and audio recordings of study telephone sessions will be stored on Duke servers.

ELIGIBILITY:
Inclusion Criteria:

* being at least 21 years of age
* a diagnosis of stage IV cancer in the past 3 years
* being able to speak/read English

Exclusion Criteria:

* visual or hearing impairment that would prevent ability to engage in the telephone session or study materials
* presence of a severe unmanaged psychiatric condition (i.e., psychotic disorder or episode) or a psychiatric condition (e.g., suicidal intent) that would contraindicate safe participation in the study as indicated by the medical chart, treating oncologist, or interactions with the medical/study staff.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-01-03 (Actual); Primary Completion 2018-09-08 (Actual); Study Completion 2018-09-08 (Actual)

PRIMARY OUTCOMES:
Feasibility as measured by study attrition which will be assessed by patients who do not complete the post-assessment. | 8 weeks
  Feasibility will be shown by no more than 20% study attrition.
Acceptability, as measured by Client Satisfaction Questionnaire 10-item version | 8 weeks
  Acceptability will be indicated by at least 80% of the participants reporting satisfaction with the CBT protocol (mean score of 7) on the CSQ
Feasibility as measured by study accrual by meeting recruitment goal | 8 weeks
  Feasibility will be shown by meeting targeted study accrual (N=35) in the 12-month study period.
Feasibility as measured by adherence to the study protocol by number of intervention sessions completed by the participant | 8 weeks
  Feasibility will be shown by adherence to at least 75% of the intervention sessions (3/4)

SECONDARY OUTCOMES:
Change in pain | Baseline and 8 weeks
  Pain will be assessed with the Brief Pain Inventory (BPI)
Change in fatigue | Baseline and 8 weeks
  Fatigue will be assessed with the PROMIS Adult Fatigue Profile Short Form.
Change in depression | Baseline and 8 weeks
  The Hospital Anxiety and Depression Scale will be used to assess distress (anxiety and depressive symptoms)
Change in Mindfulness | Baseline and 8 weeks
  Acceptance and mindfulness will be assessed using the Acceptance and Action Questionnaire-II, the most widely used measure of mechanism of change in ACT-based medical treatment studies.
Change in anxiety | Baseline and 8 weeks
  The Hospital Anxiety and Depression Scale will be used to assess distress (anxiety and depressive symptoms)
Change in Acceptance | Baseline and 8 weeks
  Acceptance and mindfulness will be assessed using the Acceptance and Action Questionnaire-II, the most widely used measure of mechanism of change in ACT-based medical treatment studies.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Plumb Vilardaga, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States